CLINICAL TRIAL: NCT05463042
Title: Effect of Intermittent Hypoxia on Balance Control During Standing and Walking in Healthy Adults
Brief Title: Intermittent Hypoxia and Balance Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Hao-Yuan Hsiao, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003081
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Intermittent Hypoxia; Normoxia
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: This is a cross-over design study that requires 2 visits (a least 1-week apart). Fifteen younger adults and 15 older adults will be recruited. Participants will be pseudo-randomly assigned to receive either intermittent hypoxia or sham during the first visit, and then switch over to receive sham or intermittent hypoxia during the 2nd visit.
Who Masked: Participant
Masking Description: Participants will not be informed about which condition (intermittent hypoxia or normoxia) they are experiencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Hypoxia (Experimental): Participants will receive intermittent hypoxia and perform balance and gait assessments before and after the intermittent hypoxia session.
  Interventions: Behavioral: Intermittent Hypoxia
- Normoxia (sham) (Sham Comparator): Participants will receive normoxia and perform balance and gait assessments before and after the normoxia session.
  Interventions: Behavioral: Normoxia (sham)

INTERVENTIONS:
Behavioral: Intermittent Hypoxia — During the intermittent hypoxia session, participants will be sitting during the entire breathing protocol. Hypoxic air will be inhaled through a mask connected to a two-way non-rebreathing valve, which will itself be connected to a 5-liter non-diffusing gas bag (Hans Rudolph, Inc, USA). The rebreathing bag will be connected to a certified medical grade gas tank containing 11% oxygen and a balance of nitrogen. The intermittent hypoxia protocol will consist of eight 4-min cycles of breathing hypoxic air interspersed with normoxic cycles breathing room air. After four min of hypoxia, participants will be switched back to breathing room air until resaturation, which takes approximately one minute. Once arterial oxygen saturation reaches baseline levels, participants will be switched back to breathing hypoxic air, beginning the next hypoxic cycle.
  Arms: Intermittent Hypoxia
Behavioral: Normoxia (sham) — During the sham condition, compressed air (21% oxygen) from a gas tank will be delivered throughout the protocol instead of 11% oxygen. Participants will not receive information about which condition (Intermittent hypoxia or sham) they are experiencing during the trials.
  Arms: Normoxia (sham)

SUMMARY:
This study aims to determine the effect of acute mild intermittent hypoxia on ankle plantarflexor muscle output during balance regulation and walking in younger and older adults. Fifteen younger adults and 15 older adults will be recruited to participate in the cross-over design study that requires 2 visits (at least 1-week apart). Participants will be pseudo-randomly assigned to receive either intermittent hypoxia or sham during the first visit, and then switch over to receive sham or intermittent hypoxia during the 2nd visit. Muscle activation patterns and kinetic and kinematics during standing and walking will be recorded before and after the intermittent hypoxia/sham. It is hypothesized that compared to the sham condition, both younger and older participants will show greater increases in ankle plantarflexor muscle activation during gait and balance assessments following intermittent hypoxia.

DETAILED DESCRIPTION:
Procedure:

This is a cross-over design study that requires 2 visits (at least 1-week apart). Fifteen younger adults and 15 older adults will be recruited. Participants will be pseudo-randomly assigned to receive either intermittent hypoxia or sham during the first visit, and then switch over to receive sham or intermittent hypoxia during the 2nd visit.

During each visit, participants will first perform Gait and Balance Assessments (PRE), followed by the Intermittent Hypoxia (or sham) protocol, and then perform Gait and Balance Assessments (POST) again. The total time is approximately 2.5 hours for each visit.

Balance and Gait Assessments The consent process and Balance and Gait Assessments will take place in BEL 530.

During Balance and Gait Assessments, participants will be asked to wear tight-fitting shorts and shirt for accurate marker positioning. Approximately 39 reflective markers will be attached to target locations on the individuals' body (the head, arms, wrists, hands, trunk, pelvis, legs and feet) according to the Vicon Full-Body Plug-In Gait Model.

A study team member will attach surface electrodes over the tibialis anterior and soleus muscles to record the muscle activation patterns with a wireless Electromyography (EMG) system (Delsys Inc., Natick, MA). Next, a study team member will assist the participant to wear a safety harness that will be attached to an overhead support beam.

For Balance Assessment, participants will stand on the treadmill with their feet shoulder-width apart. A 30-second quiet standing trial will be recorded. Next, participants will be instructed to maintain upright posture when the treadmill shifts forward or backward at unknown times (perturbed standing). The treadmill will shift approximately 3 cm. Based on our previous experiment, this distance is sufficient to trigger a response without inducing a fall. Three forward and 3 backward treadmill shifts will be delivered in a randomized order. Finally, participants will be asked to close their eyes and repeat the quiet standing and perturbed standing trials. A 10-camera Vicon Nexus motion capture system (Vicon, Oxford Metrics, UK) will be used to record whole body kinematics. Ground reaction forces under each belt will be recorded. A handrail is located on either side of the treadmill.

For Gait Assessments, participants will walk on the treadmill at their comfortable and fast walking speeds. The comfortable speed will be determined by gradually increasing the treadmill speed until the participant confirms that it reaches their comfortable regular walking speed. The fast speed will be determined by gradually increasing the treadmill speed until the participant confirms that it reaches the maximum speed that they can walk safely. A 30-second walking trial will be recorded for each speed.

Following Balance and Gait Assessment, a testing team member will escort the participant to BEL819 Clinical Exercise Physiology Laboratory to perform Intermittent Hypoxia (or sham).

Intermittent hypoxia Intermittent hypoxia will be performed in BEL819 Clinical Exercise Physiology Laboratory. Intermittent hypoxia is routinely performed in this laboratory (IRB protocols 2017090015, 2018110129, 2019070088, and 202005018). Intermittent hypoxia consisting of a limited number (5-10/day) of short (4-10 min) bouts of mild hypoxia (oxygen levels between 10-12%) leads to cumulative and sustained beneficial physiological responses. Preliminary data collected in the Clinical Exercise Physiology Laboratory show that a fraction of oxygen of 11±1% corresponds to an arterial oxygen saturation of 80±2% in middle-aged individuals. Participants will be sitting during the entire breathing protocol. Hypoxic air will be inhaled through a mask connected to a two-way non-rebreathing valve, which will itself be connected to a 5-liter non-diffusing gas bag (Hans Rudolph, Inc, USA). The rebreathing bag will be connected to a certified medical grade gas tank containing 11% oxygen and a balance of nitrogen. The intermittent hypoxia protocol will consist of eight 4-min cycles of breathing hypoxic air interspersed with normoxic cycles breathing room air. After four min of hypoxia, participants will be switched back to breathing room air until resaturation, which takes approximately one minute. Once arterial oxygen saturation reaches baseline levels, participants will be switched back to breathing hypoxic air, beginning the next hypoxic cycle. Unlike chronic hypoxic exposure, risks associated with an acute hypoxic exposure of three 4-min cycles are minimal, and no adverse events were reported during intermittent hypoxia in our participants.

During the sham condition, compressed air (21% oxygen) from a gas tank will be delivered throughout the protocol instead of 11% oxygen. Participants will not receive information about which condition (Intermittent hypoxia or sham) they are experiencing during the trials.

Pulmonary gas exchange Breath-by-breath measures of pulmonary gas exchange such as volume of oxygen and carbon dioxide, respiratory rate, tidal volume, minute ventilation and fraction of inspired oxygen will be determined from a pneumotachometer (Ultima Cardio2, MGC Diagnostics, MN, USA) throughout the intermittent hypoxia. The pneumotachometer will be mounted between the mask and the non-rebreathing valve of the breathing circuit. The pneumotachometer, mouthpiece and non-rebreathing valve will be disinfected in a 10% bleach and water solution for 60 minutes and rinse thoroughly with tap water for 5 minutes between each use. Each participant will have a face mask that will only be used by him/her.

Hemodynamics An arterial waveform obtained by finger plethysmography from the middle finger of the left hand will be continuously recorded (NOVA, Finapres Medical Systems, Amsterdam, Netherlands) during the intermittent hypoxia. Systolic, diastolic and mean arterial pressure, heart rate, stroke volume, cardiac output and total peripheral resistance will be derived from the arterial waveform, a method which has been validated against invasive measures [9]. All data will be recorded in LabChart (Powerlab, ADInstruments Inc., CO, USA) for later analysis.

Arterial oxygen saturation Arterial oxygen saturation will continuously be monitored by pulse oximetry (NOVA, Finapres Medical Systems, Amsterdam, Netherlands) throughout the intermittent hypoxia. The pulse oximeter probe will be applied to the index finger of the left hand.

Following intermittent hypoxia (or sham), a testing team member will escort the participant back to BEL530 to perform Balance and Gait Assessment. After the assessment, a testing team member will remove the electrodes and markers from the participant.

ELIGIBILITY:
Inclusion Criteria:

- Able to stand and walk for more than 5 minutes without assistance.

Exclusion Criteria:

* Have high blood pressure (above 130/90 mmHg)
* Are smokers
* Are pregnant
* Have body mass index more than 35 kg/m2
* Have a history of falls in the past 6 months
* Have a history of neuromuscular deficits that may affect gait
* Have a history of cardiovascular disease
* Have a history of diabetes or lung disease
* Are taking medication affecting the cardiovascular system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Soleus muscle activation pattern | pre (2o minutes before) and post (20 minutes after) intermittent hypoxia or sham session
  changes in peak soleus muscle EMG magnitude following perturbation onset during standing from pre to post intermittent hypoxia will be calculated
Ankle plantarflexion torque | pre (20 minutes before) and post (20 minutes after) intermittent hypoxia or sham session
  Changes in peak ankle plantarflexion torque production during walking from pre to post intermittent hypoxia will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This proposed research will include data from approximately 30 subjects regarding their walking and standing balance control mechanics. Muscle activation patterns, body movement, and force production data will be recorded. Only de-identified data will be shared for research purposes.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available following the completion of data analyses for 10 years.

REFERENCES:
- [Background] Mateika JH, El-Chami M, Shaheen D, and Ivers B. Intermittent hypoxia: a low-risk research tool with therapeutic value in humans. J Appl Physiol (1985). 2015. 118(5): 520-32. Meerson F, Pozharov V, and Minyailenko T. Superresistance against hypoxia after preliminary adaptation to repeated stress. J Appl Physiol (1985). 1994. 76(5): 1856-61. Neubauer JA. Invited review: Physiological and pathophysiological responses to intermittent hypoxia. J Appl Physiol (1985). 2001. 90(4): 1593-9. Casey DP, Shepherd JR, and Joyner MJ. Sex and vasodilator responses to hypoxia at rest and during exercise. J Appl Physiol (1985). 2014. 116(7): 927-36. Casey DP, Walker BG, Curry TB, and Joyner MJ. Ageing reduces the compensatory vasodilatation during hypoxic exercise: the role of nitric oxide. J Physiol. 2011. 589(Pt 6): 1477-88. Jarrard CP, Nagel MJ, Stray-Gundersen S, Tanaka H, and Lalande S. Hypoxic preconditioning attenuates ischemia-reperfusion injury in young healthy adults. J Appl Physiol (1985). 2021. 130(3): 846-852. Nagel MJ, Jarrard CP, and Lalande S. Effect of a Single Session of Intermittent Hypoxia on Erythropoietin and Oxygen-Carrying Capacity. Int J Environ Res Public Health. 2020. 17(19). Wojan F, Stray-Gundersen S, Nagel MJ, and Lalande S. Short exposure to intermittent hypoxia increases erythropoietin levels in healthy individuals. J Appl Physiol (1985). 2021. 130(6): 1955-1960. Wesseling KH, Jansen JR, Settels JJ, and Schreuder JJ. Computation of aortic flow from pressure in humans using a nonlinear, three-element model. J Appl Physiol (1985). 1993. 74(5): 2566-73.